CLINICAL TRIAL: NCT07263386
Title: A Phase II, Multicenter, Randomized, Controlled Clinical Study Comparing the Efficacy and Safety of Sintilimab Plus SOX Versus SOX Alone as Adjuvant Therapy for PD-L1-Positive, Stage pN3 Gastric Cancer
Acronym: ARTEMIS-GC3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-859
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Gastric Adenocarcinoma
Keywords: PD-1 inhibitor; adjuvant therapy; Sintilimab; Gastric Adenocarcinoma
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab + SOX (Active Comparator): Patients will first receive 6 to 8 cycles of treatment with sintilimab + SOX; sintilimab will subsequently be continued as maintenance therapy for up to one year.
  Interventions: Drug: Sintilimab; Drug: SOX Chemotherapy
- SOX (Active Comparator): Patients will receive 6 to 8 cycles of treatment with SOX
  Interventions: Drug: SOX Chemotherapy

INTERVENTIONS:
Drug: Sintilimab — For patients with body weight < 60 kg, the dose is 3 mg/kg, administered via intravenous infusion (i.v.gtt.) on Day 1; for patients with body weight ≥ 60 kg, a fixed dose of 200 mg is administered via intravenous infusion (i.v.gtt.) on Day 1. The treatment is repeated every 21 days.
  Arms: Sintilimab + SOX
Drug: SOX Chemotherapy — S-1: 40 mg/m², oral administration (p.o.), twice daily (b.i.d.), on Days 1 to 14; repeated every 21 days.
  Oxaliplatin: 130 mg/m², intravenous infusion (i.v.gtt.), on Day 1; repeated every 21 days.

SUMMARY:
This study intends to enroll gastric cancer patients who are PD-L1 positive and pathologically confirmed as Stage N3. Enrolled patients will be randomly assigned to receive either standard adjuvant SOX regimen or SOX regimen combined with sintilimab. The objective of the study is to determine whether adding a PD-1 inhibitor to postoperative chemotherapy can improve the Disease-Free Survival (DFS) rate in patients with Stage N3 gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent form prior to the initiation of any study-related procedures.
* Aged between 18 and 75 years.
* Have undergone radical resection with D2 or wider lymph node dissection and achieved R0 resection status.
* No prior systemic anti-tumor treatment (i.e., neoadjuvant therapy) before surgery.
* Histopathologically confirmed gastric adenocarcinoma.
* Pathological stage classified as TxN3M0 according to the 8th edition of the AJCC Cancer Staging Manual.
* PD-L1 Combined Positive Score (CPS) ≥ 1.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Expected survival time ≥ 6 months.
* Adequate organ function, with subjects meeting the following laboratory criteria before enrollment:

Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L without the use of granulocyte colony-stimulating factor (G-CSF) within the past 14 days.

Platelet count ≥ 100×10⁹/L without blood transfusion within the past 14 days. Hemoglobin > 9 g/dL without blood transfusion or use of erythropoietin within the past 14 days.

Total bilirubin ≤ 1.5×Upper Limit of Normal (ULN); subjects with total bilirubin > 1.5×ULN but direct bilirubin ≤ ULN are also eligible.

Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5×ULN. Serum creatinine ≤ 1.5×ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min.

Adequate coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5×ULN.

Normal thyroid function, defined as Thyroid-Stimulating Hormone (TSH) within the normal range. Subjects with baseline TSH outside the normal range are eligible if total T3 (or free T3, FT3) and free T4 (FT4) are within the normal range.

Myocardial enzyme profile within the normal range (subjects with isolated laboratory abnormalities deemed clinically insignificant by the investigator are also eligible).

* For female subjects of childbearing potential, a negative urine or serum pregnancy test must be obtained within 3 days before the first administration of the study drug (Cycle 1, Day 1). A blood pregnancy test is required if the urine pregnancy test result is inconclusive. Non-childbearing potential is defined as postmenopausal for at least 1 year, or having undergone surgical sterilization or hysterectomy.
* All subjects (male and female) at risk of conception must use contraceptive methods with a yearly failure rate of less than 1% throughout the treatment period and until 120 days after the last administration of the study drug (or 180 days after the last administration of chemotherapy drugs).

Exclusion Criteria:

* Pathologically confirmed as squamous cell carcinoma, adenosquamous carcinoma, undifferentiated carcinoma, neuroendocrine tumor, or gastrointestinal stromal tumor (mixed carcinoma with adenocarcinoma component > 80% is eligible for enrollment).
* Diagnosis of malignant diseases other than gastric cancer within 5 years before the first dose administration (excluding radically treated basal cell carcinoma of the skin, cutaneous squamous cell carcinoma, differentiated thyroid cancer, and/or radically resected carcinoma in situ).
* Currently participating in therapeutic clinical research, or having received other study drugs within 4 weeks before the first dose administration.
* Previous receipt of the following therapies: anti-PD-1, anti-PD-L1, or drugs targeting other stimulatory or co-inhibitory T-cell receptors (including but not limited to CTLA-4, OX-40, CD137, etc.).
* Receipt of Chinese patent medicines with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural effusion) via systemic treatment within 2 weeks before the first dose administration.
* History of active autoimmune diseases requiring systemic treatment (e.g., disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years before the first dose administration. Replacement therapies (e.g., thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic treatment.
* Receipt of systemic glucocorticoid therapy (excluding nasal, inhaled, or other forms of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first dose administration of the study; Note: - - Use of physiological doses of glucocorticoids (≤ 10 mg/day prednisone or equivalent drugs) is allowed.
* Known history of allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* Known history of allergy to drugs used in this study.
* Failure to fully recover from toxicity and/or complications caused by any intervention before the start of treatment (i.e., ≤ Grade 1 or return to baseline, excluding fatigue or alopecia).
* Known history of human immunodeficiency virus (HIV) infection (i.e., positive HIV 1/2 antibodies).
* Untreated active hepatitis B (defined as positive HBsAg with HBV-DNA copy number exceeding the upper limit of normal value of the laboratory in the research center); Note: Hepatitis B subjects meeting the following criteria are also eligible: HBV viral load < 1000 copies/ml (200 IU/ml) before the first dose administration, and subjects should receive anti-HBV treatment during the entire study chemotherapy period to avoid viral reactivation. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and negative HBV viral load, prophylactic anti-HBV treatment is not required, but close monitoring of viral reactivation is necessary.
* Subjects with active HCV infection (positive HCV antibody and HCV-RNA level above the lower limit of detection).
* Receipt of live vaccines within 30 days before the first dose administration (Cycle 1, Day 1); Note: Receipt of inactivated influenza vaccines via injection within 30 days before the first dose administration is allowed, but intranasal attenuated live influenza vaccines are not allowed.
* Pregnant or lactating women.
* Presence of any severe or uncontrolled systemic diseases, such as:

Significant and poorly controlled abnormalities in rhythm, conduction, or morphology on resting electrocardiogram, such as complete left bundle branch block, second-degree or higher atrioventricular block, ventricular arrhythmia, or atrial fibrillation.

Unstable angina pectoris, congestive heart failure, or chronic heart failure with New York Heart Association (NYHA) classification ≥ Grade 2.

Any arterial thrombosis, embolism, or ischemia (e.g., myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack) within 6 months before enrollment.

Poorly controlled blood pressure (systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg despite medication).

History of non-infectious pneumonia requiring glucocorticoid treatment within 1 year before the first dose administration, or current clinically active interstitial lung disease.

Active pulmonary tuberculosis. Presence of active or uncontrolled infection requiring systemic treatment. Presence of clinically active diverticulitis, abdominal abscess, or gastrointestinal obstruction.

Liver diseases such as cirrhosis, decompensated liver disease, and acute or chronic active hepatitis.

Poorly controlled diabetes mellitus (fasting blood glucose (FBG) > 10 mmol/L). Urinalysis indicating urine protein ≥ ++, and confirmed 24-hour urine protein > 1.0 g.

Patients with mental disorders who are unable to cooperate with treatment.

- Presence of medical history, evidence of disease, treatment, or abnormal laboratory test results that may interfere with study results, prevent the subject from completing the study, or other circumstances deemed unsuitable for enrollment by the investigator, or other potential risks deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | 3 years
  Defined from the date of completion of curative-intent treatment (e.g., surgery, adjuvant chemotherapy) to the date of first documentation of disease recurrence (e.g., tumor relapse, metastasis) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Defined from date of recruit to date of first documentation of death from any cause or censored at the date of the last follow-up.
Incidence rate of adverse events (AEs) | 3 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Serious adverse events (SAE) | 3 years
  Serious adverse events (SAE) is defined as either death, life-threatening, or Permanent or severe disability/incapacity.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China